CLINICAL TRIAL: NCT04202822
Title: Early Healing of Oral Soft Tissues: a Clinical and Biomolecular Analysis Part I - Gene Expression and Cellular Behaviour 24-hours After Injury
Brief Title: Early Healing of Oral Soft Tissues: a Clinical and Biomolecular Analysis. Part I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5315 Prot 2018/19
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Wound Surgical; Wound Heal; Oral Soft Tissue Conditions
Keywords: real-time polymerase chain reaction; early wound healing; gingiva; oral mucosa
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsies (Other): Oral soft tissues biopsies (alveolar mucosa, buccal gingiva, and palatal tissue) at T0 and T24
  Interventions: Other: Oral soft tissues biopsies

INTERVENTIONS:
Other: Oral soft tissues biopsies — Oral soft tissues biopsies (alveolar mucosa, buccal gingiva, and palatal tissue) will be harvested by the examiner at the time of the surgery (immediately before to start the surgical procedure -T0) and 24 hours after surgery (T24) at the level of the vertical released incisions (VRIs) with a biopsy punch with plunger of 2.0 mm diameter.

SUMMARY:
The purpose of the present study is to observe and compare -through a biomolecular analysis- the differences in the gene expression and cellular behavior in the early wound healing process -24 hours after injury- between the following three oral tissues: alveolar mucosa, buccal gingiva and palatal tissue.

The main hypothesis is that there is a difference in the gene expression and in the cellular behaviour between the three oral tissues studied and this difference can be observed at 24 hours post-injury.

DETAILED DESCRIPTION:
The wound healing is an extremely complex process. It has been observed that oral wounds mechanisms present special features. In fact, mucosal wounds demonstrated accelerated healing compared to cutaneous wounds.

Numerous comparative studies have described important differences of cellular behavior and genes expression between oral mucosal and dermal tissues. Moreover, it has been observed that the behavior of the cells is autonomous, i.e., that greatest differences seen in the genomic response after injury in skin and mucosa are derived, in part, from intrinsic differences in the genetic regulation of the cells at each site. Also, it is important to highlight the fact that it has been observed that the cellular response after wound is early, showing the first and greatest changes at 12-24 hours post injury. Moreover, a recent study has been raised the possibility of that the transcriptional regulatory networks responsible for the accelerated healing in oral mucosa are already present in the unwounded state.

In the oral mucosal tissues, the mechanisms underlying scar-less wound healing have been studied. Most studies have focused on the cellular characteristics and the molecular expression as growing factors, inflammatory mediators, etc., and have evaluated the process in later periods.

Therefore, while the biomolecular basis of the differences in oral mucosal and dermal tissues wound healing have been described, this is less well understood in the different oral soft tissue wounds.

The following points must be considered:

* The differences in the wound healing between mucosal and dermal tissues have been extensively studied through biomolecular analysis.
* The behavior of the cells is autonomous.
* The changes in the wound healing have been observed after 12-24 hours post-injury.
* The transcriptional regulatory networks responsible for the accelerated healing in oral mucosa could already be present in the unwounded state.
* The differences in the wound healing between the different oral soft tissues (alveolar mucosa, buccal gingiva and palatal tissue) has not been studied from a biomolecular point of view; however, differences in the clinical behavior and response between these three oral tissues has been reported.

The main questions are:

1. Twenty-four hours after injury: Are there differences in the gene expression and cellular behaviour between the three studied tissues?
2. The transcriptional regulatory networks responsible for the accelerated oral tissues healing:

   * Are presents in the unwounded state?
   * Are differences between the three studied oral tissues?

Deepen the knowledge in the early wound healing process of these tissues and the difference between them -evaluating the genes expression and the behavior of the cells- could allow the generation of new approaches to improve the healing of oral wounds.

ELIGIBILITY:
Inclusion Criteria:

* patients that required periodontal surgery;
* patients age between 30-60 years;
* patients with full mouth plaque score and full mouth bleeding score < 15%;
* patients with a good general healthy status;
* patients without any medicaments or drug consumption that can affect the healing process;
* non-smoking patients.

Exclusion Criteria:

* patients in pregnancy;
* patients in lactation period;
* patients with consumption of antibiotics or anti-inflammatory drugs in the previous six months;
* patients with systemic diseases.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Changes from baseline fold regulation wound healing related genes at 24 hours | Baseline (T0) and 24 hours after surgery (T24)
  Total RNA from biopsies or cell cultures was extracted using TRIzol reagent Quantitative real-time PCR (qRT-PCR) cDNA was generated and cDNA obtained were used for amplification of wound healing related genes using the appropriate TaqMan gene expression assay kits.

SECONDARY OUTCOMES:
Clinical evaluation of early wound healing | 24 hours and 1 week after surgery
  Assessed with a clinical index (EHS- Early wound healing score). This score assessed clinical signs of re-epithelialization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Since complete wound epithelialization was the main outcome, the CSR score was weighted to be 60% of the total final score. Accordingly, a score of 0, 3, or 6 points was possible for the assessment of CSR, whereas scores of 0, 1, or 2 points were possible for CSH and CSI. Higher values indicated better healing. Accordingly, the score for ideal early wound healing was 10.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD,DDS,MS, Study Director — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillofacial Sciences. Section of Periodontics.Sapienza, University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eming SA, Martin P, Tomic-Canic M. Wound repair and regeneration: mechanisms, signaling, and translation. Sci Transl Med. 2014 Dec 3;6(265):265sr6. doi: 10.1126/scitranslmed.3009337. PMID 25473038
- [Background] Bartold PM, McCulloch CA, Narayanan AS, Pitaru S. Tissue engineering: a new paradigm for periodontal regeneration based on molecular and cell biology. Periodontol 2000. 2000 Oct;24:253-69. doi: 10.1034/j.1600-0757.2000.2240113.x. No abstract available. PMID 11276871
- [Background] Szpaderska AM, Walsh CG, Steinberg MJ, DiPietro LA. Distinct patterns of angiogenesis in oral and skin wounds. J Dent Res. 2005 Apr;84(4):309-14. doi: 10.1177/154405910508400403. PMID 15790734
- [Background] Warburton G, Nares S, Angelov N, Brahim JS, Dionne RA, Wahl SM. Transcriptional events in a clinical model of oral mucosal tissue injury and repair. Wound Repair Regen. 2005 Jan-Feb;13(1):19-26. doi: 10.1111/j.1067-1927.2005.130104.x. PMID 15659033
- [Background] Wong JW, Gallant-Behm C, Wiebe C, Mak K, Hart DA, Larjava H, Hakkinen L. Wound healing in oral mucosa results in reduced scar formation as compared with skin: evidence from the red Duroc pig model and humans. Wound Repair Regen. 2009 Sep-Oct;17(5):717-29. doi: 10.1111/j.1524-475X.2009.00531.x. PMID 19769724
- [Background] Mak K, Manji A, Gallant-Behm C, Wiebe C, Hart DA, Larjava H, Hakkinen L. Scarless healing of oral mucosa is characterized by faster resolution of inflammation and control of myofibroblast action compared to skin wounds in the red Duroc pig model. J Dermatol Sci. 2009 Dec;56(3):168-80. doi: 10.1016/j.jdermsci.2009.09.005. Epub 2009 Oct 24. PMID 19854029
- [Background] Roy S, Khanna S, Rink C, Biswas S, Sen CK. Characterization of the acute temporal changes in excisional murine cutaneous wound inflammation by screening of the wound-edge transcriptome. Physiol Genomics. 2008 Jul 15;34(2):162-84. doi: 10.1152/physiolgenomics.00045.2008. Epub 2008 May 6. PMID 18460641
- [Background] Chen W, Fu X, Ge S, Sun T, Zhou G, Han B, Li H, Sheng Z. Profiling of genes differentially expressed in a rat of early and later gestational ages with high-density oligonucleotide DNA array. Wound Repair Regen. 2007 Jan-Feb;15(1):147-55. doi: 10.1111/j.1524-475X.2006.00195.x. PMID 17244330
- [Background] Iglesias-Bartolome R, Uchiyama A, Molinolo AA, Abusleme L, Brooks SR, Callejas-Valera JL, Edwards D, Doci C, Asselin-Labat ML, Onaitis MW, Moutsopoulos NM, Gutkind JS, Morasso MI. Transcriptional signature primes human oral mucosa for rapid wound healing. Sci Transl Med. 2018 Jul 25;10(451):eaap8798. doi: 10.1126/scitranslmed.aap8798. PMID 30045979
- [Background] Wang Y, Tatakis DN. Human gingiva transcriptome during wound healing. J Clin Periodontol. 2017 Apr;44(4):394-402. doi: 10.1111/jcpe.12669. Epub 2017 Feb 11. PMID 28005267
- [Background] Kantarci A, Black SA, Xydas CE, Murawel P, Uchida Y, Yucekal-Tuncer B, Atilla G, Emingil G, Uzel MI, Lee A, Firatli E, Sheff M, Hasturk H, Van Dyke TE, Trackman PC. Epithelial and connective tissue cell CTGF/CCN2 expression in gingival fibrosis. J Pathol. 2006 Sep;210(1):59-66. doi: 10.1002/path.2000. PMID 16841303
- [Background] Vescarelli E, Pilloni A, Dominici F, Pontecorvi P, Angeloni A, Polimeni A, Ceccarelli S, Marchese C. Autophagy activation is required for myofibroblast differentiation during healing of oral mucosa. J Clin Periodontol. 2017 Oct;44(10):1039-1050. doi: 10.1111/jcpe.12767. Epub 2017 Aug 25. PMID 28646601
- [Background] Marini L, Rojas MA, Sahrmann P, Aghazada R, Pilloni A. Early Wound Healing Score: a system to evaluate the early healing of periodontal soft tissue wounds. J Periodontal Implant Sci. 2018 Oct 24;48(5):274-283. doi: 10.5051/jpis.2018.48.5.274. eCollection 2018 Oct. PMID 30405935
- [Derived] Rojas MA, Ceccarelli S, Gerini G, Vescarelli E, Marini L, Marchese C, Pilloni A. Gene expression profiles of oral soft tissue-derived fibroblast from healing wounds: correlation with clinical outcome, autophagy activation and fibrotic markers expression. J Clin Periodontol. 2021 May;48(5):705-720. doi: 10.1111/jcpe.13439. Epub 2021 Feb 17. PMID 33527447